CLINICAL TRIAL: NCT01296685
Title: Clinical Evaluation of Air Handling in Baby fx Oxygenator With Integrated Arterial Filter Versus Baby rx Oxygenator With Non Integrated Arterial Line Filter
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Dr. Al Tmimmi, University Hospitals Leuven
Other Study IDs: S 52937
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-02

CONDITIONS: Cardiovascular Surgical Procedure
Keywords: cardiovascular surgical procedure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- oxygenator with arterial filter
- arterial filter

SUMMARY:
The goal of the study is the evaluation of the air handling of a "new" type of oxygenator versus the standard model. The new type has an integrated arterial filter. The standard model has a non integrated arterial line filter. If the air handling is as effective/ better than in the standard model this can lead to reduction of cardiopulmonary bypass circuits with their initiation of systemic inflammatory response and improve cardiopulmonary bypass safety.

ELIGIBILITY:
Inclusion Criteria:

* All children with body surface area between 0.25 and 0.5 m² who need cardiac surgery with cardiopulmonary bypass.

Exclusion Criteria:

* Urgent and norwood procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All children with body surface area between 0.25 and 0.5 m² who need cardiac surgery with cardiopulmonary bypass. Urgent and norwood procedures are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-03

CONTACTS AND LOCATIONS:
Overall Officials: Layth Al Tmimi, Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven